CLINICAL TRIAL: NCT05095805
Title: Weight-bearing Training Exercise May Improve Loading of Trans-tibial Prosthesis and Functional Gait
Brief Title: Weight-bearing Exercise for Trans-tibial Amputees
Acronym: Prototest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Rehabilitation Institute, Republic of Slovenia (Other)
Collaborators: Slovenian Research Agency (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URIS202102
Record Dates: First submitted 2021-10-14; First posted 2021-10-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Amputation
Keywords: trans-tibial prosthesis; weight-bearing; balance; centre of pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): additional weight-bearing exercise
  Interventions: Behavioral: additional weight-bearing exercise
- Control group (Active Comparator): standard weight-bearing exercise
  Interventions: Behavioral: standard weight-bearing exercise

INTERVENTIONS:
Behavioral: additional weight-bearing exercise — Nintendo Wii Balance Board, real-time visual feedback, weight-bearing assessment by center of pressure
  Arms: Test group
Behavioral: standard weight-bearing exercise — conventional training for fitting of initial prosthesis
  Arms: Control group

SUMMARY:
A simple weight-bearing exercise has been designed using off-the-shelves devices (Nintendo Wii Balance Board) and centre of pressure (COP) analysis software (Python) for trans-tibial amputees receiving their first prosthesis. A pilot randomised control study will be conducted to check the progress with weight-bearing training using COP-based objective measures. Additionally, gait and functional task performance will be assessed by means of clinical test. Participants will be divided into 2 groups: test group (performing additional weight-bearing exercises) and control group (receiving only conventional training for fitting of initial prosthesis).

DETAILED DESCRIPTION:
Each patient meeting the inclusion criteria will be randomised to either the test group or the control group. The patients will perform ten training sessions with the initial prosthesis, each session lasting for about 30 minutes, within the period of two weeks. They will be assessed at baseline and after the training program.

ELIGIBILITY:
Inclusion Criteria:

* trans-tibial amputation,
* fitted with first trans-tibial prosthesis,
* independent mobility for 50m with or without assistive aid,
* Functional Independence Measure (FIM) Stairs locomotion scale ≥ 5,
* ability to follow the instructions, Mini Mental State Examination (MMSE) > 25,
* no severe visual problems, ble to see computer screen,
* willing to participate.

Exclusion Criteria:

* bilateral lower limb amputation or any other level of unilateral lower limb amputation,
* not candidates for prosthetic fitting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in centre of pressure (COP) from baseline | Assessment at baseline and after two weeks
  Calculation of COP (transversal plane, symmetry index, lateral, sagittal directions) from 4 pressure sensors built into the balance board
Change in weight distribution in quiet standing | Assessment at baseline and after two weeks
  COP assessment for 20s of quiet standing

SECONDARY OUTCOMES:
Change in 10m walk test | Assessment at baseline and after two weeks
Change in L-test | Assessment at baseline and after two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Helena Burger, MD, PhD, Study Chair — University Rehabilitation Institute, Republic of Slovenia
Locations (1):
- University Rehabilitation Institute, Republic of Slovenia, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No